CLINICAL TRIAL: NCT06804694
Title: Technology-Enabled Collaborative Care for Young Adults With Type-1 Diabetes and Diabetes Distress (TECCT1D3): Feasibility Trial of a Co-designed Intervention
Brief Title: Technology-Enabled Collaborative Care for Young Adults With Type 1 Diabetes and Diabetes Distress: A Feasibility Trial
Acronym: TECC-T1D3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brain Canada (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Peter Selby, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/065
Record Dates: First submitted 2025-01-06; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes (T1D); Diabetes Distress
Keywords: Type 1 Diabetes; TECC model; Diabetes Distress; Technology-enabled Care; Young adults with T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coaching Intervention (TECC-T1D3 Program) (Experimental): Participants will complete a 12-weeks, virtual, TECC-T1D3 program, delivered through an omnichannel, patient-centered approach, which may include WebEx, phone calls, or text messaging. The participants will complete weekly coaching sessions with the health coach and is indirectly supported by a virtual care team comprised of mental health and T1D experts as well as peer support.
  Interventions: Behavioral: TECC-T1D3 Program
- Education Intervention (Active Comparator): Participants will receive a low-intensity, education-focused intervention consisting of 10 automated emails over 12 weeks, providing generalized educational messages with links to resources for mental health support and well-being for individuals living with T1D.
  Interventions: Other: Education Intervention

INTERVENTIONS:
Behavioral: TECC-T1D3 Program — The TECC-T1D3 program is a twelve-week virtual care intervention designed to support individuals with Type 1 Diabetes (T1D) and Diabetes Distress. The program includes a health coach (HC) and a virtual care team (VCT) of T1D, mental health experts and peer support, offering comprehensive care through various communication channels, including WebEx, phone calls, and text messaging. The program aims to: i. Provide T1D specific mental health and wellbeing support, ii. Provide guidance on how to communicate with others about T1D, manage stigma and ask for help with diabetes management and iii. Facilitate connections with T1D communities. Participants can choose topics of discussion based on their needs and will be directly supported by the HC and indirectly monitored by VCT.
  Arms: Coaching Intervention (TECC-T1D3 Program)
Other: Education Intervention — The Education Intervention is a low-intensity, education-focused intervention consisting of 10 automated emails over 12 weeks, providing generalized educational messages with links to resources for mental health support and well-being for individuals living with T1D.
  Arms: Education Intervention

SUMMARY:
The goal of the study is to evaluate the acceptability and feasibility of a co-designed, Technology-Enabled Collaborative Care for Young Adults with Type-1 Diabetes and Diabetes Distress (TECC-T1D3) program. Through this program, the investigators aim to deliver a collaborative care intervention, featuring a health coach and a virtual care team, designed to help participants manage mental health and overall wellbeing.

DETAILED DESCRIPTION:
A total of 60 young adults with Type 1 Diabetes (T1D) will be enrolled in the study. Participants will be randomly allocated to either a coaching intervention or an education intervention for 12 weeks. During the 12-week program, participants in the coaching intervention will take part in 8-10 sessions with a health coach, where experiences living with diabetes and goals related to diabetes management, communication with a support system, and overall wellbeing will be discussed. Participants in the education intervention will receive generalized educational messages about diabetes and diabetes distress exclusively via automated emails. Before and after the program, participants will complete surveys to provide an understanding of how diabetes and diabetes-related distress are being managed. After completing the respective interventions, participants will have a one-on-one interview with the research team to discuss their experience with the program and potential areas for improvement.

The goal of the program is to enhance the quality of life for young adults with T1D who experience significant emotional burdens associated with the condition. The study addresses a critical research gap by integrating mental health support with diabetes management, a need historically underserved in healthcare settings. By developing a structured mental health intervention that is accessible and scalable, the study addresses the need for a model of whole-person care that incorporates psychological aspects as part of standard diabetes management. The model of care and findings could potentially be applied to other chronic conditions, broadening the impact of the study beyond diabetes to other areas of chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

* Young adult (age 18-29 years)
* Resident of Ontario
* Living with a self-reported diagnosis of T1D of at least 1 year
* Individual is community-living (people who live independently in the community and are not residing in a setting that provide institutional care or support)

Exclusion Criteria:

* Unable to participate in English language
* Unable to participate via telephone or web-conferencing

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment Rate (Both Arms) | Through the study completion, an average of 6 months
  The primary outcome in this study is feasibility specifically focusing on process outcomes. This includes assessing recruitment number.
Feasibility - Engagement Rate (Both Arms) | From consent to randomization throughout the study (average of 6 months)
  The primary outcome in this study is feasibility, specifically focusing on process outcomes. This includes percentage of consented participants who proceed to randomization.
Feasibility - Completion of Study Assessments (Both Arms) | Up to 12-weeks
  Coaching Intervention: Participants attending a minimum of 8 sessions out of a possible maximum of 10 sessions Education Intervention: Participants opening a minimum of 8 emails out of the 10 emails
Acceptability - Qualitative (Both Arms) | Within two weeks post-intervention, after completing the 12-weeks program
  Participants' perceptions, experiences, and satisfaction with the intervention assessed through post-intervention interviews. Interviews will explore perceived impact on health, motivation, and suggestions for improvement.
Delivery of the Digital Intervention - Number of Sessions Completed (Coaching Intervention only) | Up to 12-weeks
  • The number of sessions completed.
Delivery of the Digital Intervention - Mode of Interaction (Coaching Intervention only) | Up to 12-weeks
  Measurement include:
  • Number of interaction categorized by the mode of delivery (web-conference, telephone or text message).
Delivery of Digital Intervention - Time Spent per Session (Coaching Intervention only) | Up to 12-weeks
  • Average time spent by health coach per interaction/session with participants in minutes.

SECONDARY OUTCOMES:
Quality of Life (Both Arms) | Baseline (Week 1) and Post-Intervention (Week 12)
  the European Quality of Life - 5 Dimensions, 5 Levels (EQ-5D-5L) scale: This measure will assess overall well-being and satisfaction with life among participants. The scale evaluates five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity.
  Unit of Measure: EQ-5D-5L index score. Minimum Value: 0 (the worst possible health state). Maximum Value: 100 (the best possible health state). Interpretation: Higher scores indicate better health-related quality of life.
Self-efficacy (Both Arms) | Baseline (Week 1) and Post-Intervention (Week 12)
  Diabetes Empowerment Scale - Short Form (DES-SF) Scale:
  This measure will evaluate participants' beliefs in their ability to effectively manage their diabetes and related challenges.
  Minimum Value: 1 (low self-efficacy). Maximum Value: 5 (high self-efficacy). Interpretation: Higher scores indicate greater self-efficacy in managing diabetes.
Diabetes Distress (Both Arms) | Baseline (Week 1) and Post-Intervention (Week 12)
  Type 1 Diabetes Distress Assessment (T1DDAS) Scale: This scale evaluates ten distinct sources of diabetes-related distress. Each source is scored individually by averaging the responses to relevant items.
  Sources: Financial Worries, Interpersonal Challenges, Management Difficulties, Shame, Hypoglycemia Concerns, Healthcare Quality, Lack of Diabetes Resources, Technology Challenges, Burden to Others, Worries About Complications.
  Minimum Value: 1 (no distress). Maximum Value: 5 (highest distress). Interpretation: Higher scores indicate a greater impact of the source on diabetes distress.
Diabetes Distress (Both Arms) | Baseline (Week 1) and Post-Intervention (Week 12)
  Problem Areas in Diabetes Scale (PAID-5) Score: This will measure the level of emotional distress and burden associated with living with Type 1 Diabetes.
  Minimum Value: 0 (no distress). Maximum Value: 20 (high distress). Interpretation: Higher scores indicate greater levels of emotional distress related to diabetes.
Self-reported HbA1C Levels (Both Arms) | Baseline (Week 1) and Post-Intervention (Week 12)
  This measure assesses blood sugar control over the past 2-3 months. Participants can choose to self-report and collection of this data will be optional.
Connectedness to Care (Both Arms) | Baseline (Week 1) and Post-Intervention (Week 12)
  This measure will assess participants' perceptions of their connection to their diabetes care and peer support using a series of 5-point Likert scale questions regarding their care and support experiences.
  Scale Values:
  1. = Strongly Agree
  2. = Agree
  3. = Neither Agree nor Disagree
  4. = Disagree
  5. = Strongly Disagree
  Minimum Value: 1 (strongest sense of connectedness). Maximum Value: 5 (lowest sense of connectedness).
  Interpretation: Lower average scores indicate a stronger sense of belonging and engagement with the T1D community.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitmore C, Mangialardi N, Saiva A, Cafazzo JA, McQuire T, Mytkolli L, St John A, Senior P, Sherifali D, Strudwick G, Selby P. Evaluating the feasibility of a co-designed technology-enabled, collaborative care program for young adults with type 1 diabetes and diabetes distress: A protocol. Digit Health. 2025 Jul 29;11:20552076251365134. doi: 10.1177/20552076251365134. eCollection 2025 Jan-Dec. PMID 40755960